CLINICAL TRIAL: NCT02601729
Title: Clinical Impact of RT-CGM Reimbursement in Belgium: a Multicenter Real-life Observational Study
Brief Title: Reimbursement Study of Continuous Glucose Monitoring in Belgium
Acronym: RESCUE
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, prof. Pieter Gillard, Prof. Dr. Pieter Gillard, KU Leuven
Other Study IDs: CGM-RESCUE
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Diabetes, Type 1
Keywords: Type 1 diabetes; real-time continuous glucose monitoring; observational study; insulin pump; Belgium
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RT-CGM population: Prospective data collection during standardized clinical follow-up and from filled out questionnaires.
- Pump only population: Retrospective data collection on demographic and clinical characteristics.

SUMMARY:
Type 1 diabetes mellitus (T1DM) is an autoimmune disease caused by an immune mediated destruction of the pancreatic β-cells. Once the pancreas has been depleted of a critical mass of β-cells the need for exogenous insulin therapy emerges. Several methods exist to administer insulin. An alternative way to administer insulin is by means of continuous subcutaneous insulin infusions (CSII) or insulin-pump therapy.The frequent execution of self-monitoring of blood glucose (SMBG) accomplished by a capillary finger-stick test is essential in the management of diabetes, but this is very limited and also lacks information about rising or falling trends in the actual glycaemia. A solution for this is the use of a Real-Time Continuous Glucose Monitoring (RT-CGM) device. Contrary to SMBG, RT-CGM measures glycaemia 24 hours a day, provides information about glucose direction and rate of change during multiple days a week. Since September 2014, RT-CGM is reimbursed in Belgium for a selected group of type 1 diabetic patients by means of a so-called "CGM convention". The main objective of the study is to evaluate the impact of real time continuous glucose monitoring reimbursement on real-life clinical care parameters of type 1 diabetic patients in Belgium after 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T1DM included in the RT-CGM reimbursement system and followed in one of 17 diabetes centers.

Exclusion Criteria:

* Patients who are not included in the RT-CGM reimbursement system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Selected group of type 1 diabetic patients by means of a so-called "CGM convention". In order to be a candidate for reimbursement, patients have to be on an insulin pump and use their RT-CGM device for more than 70 % of the time (see www.riziv.be, Nota CGV 2014/228). Reimbursement via the RT-CGM reimbursement system has been granted for an initial period of three years. As part of the requirements of the current reimbursement system, the Belgian health care authorities demanded for an evaluation after 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2014-09; Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Evolution over time of HbA1c | between 12 months before and 24 months after start RT-CGM

SECONDARY OUTCOMES:
The number of hospitalizations because of hypoglycemia and/or ketoacidosis | between 12 months before and 24 months after start RT-CGM
The number of severe hypoglycemic events | between 12 months before and 24 months after start RT-CGM
The number of hypoglycemic coma | between 12 months before and 24 months after start RT-CGM
The number of hypoglycemia with seizure | between 12 months before and 24 months after start RT-CGM
The number of hypoglycemia with need of glucagon | between 12 months before and 24 months after start RT-CGM
The number of hypoglycemic events needing help from ambulance personnel | between 12 months before and 24 months after start RT-CGM
Change in utilization of RT-CGM (= % use of RT-CGM) | between 12 months before and 24 months after start RT-CGM
Number of days absent from on work or school | between 12 months before and 24 months after start RT-CGM
Quality of life measured by the Short Form Health Survey 36-item (SF-36) version 2 questionnaire for adults | between start of RT-CGM and 24 months after start RT-CGM
  Quality of life measured by the Short Form Health Survey 36-item (SF-36) version 2 questionnaire (scale: 0 (low quality of life) - 100 (high quality of life))
Fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, worry for adults | between start of RT-CGM and 24 months after start RT-CGM
  Fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, worry (scale: 0 (not worried) - 52 (very worried))
Distress due to diabetes measured by the Problem Areas In Diabetes survey, short form (PAID-SF) questionnaire for adults | between start of RT-CGM and 24 months after start RT-CGM
  Distress due to diabetes measured by the Problem Areas In Diabetes survey, short form (PAID-SF) questionnaire (scale: 0 (no distress) - 20 (very distressed))
Quality of life measured by the Diabetes Quality of Life for Youth for children | between start of RT-CGM and 24 months after start RT-CGM
  Quality of life measured by the Diabetes Quality of Life for Youth

REFERENCES:
- [Derived] De Meulemeester J, Charleer S, Visser MM, De Block C, Mathieu C, Gillard P. The association of chronic complications with time in tight range and time in range in people with type 1 diabetes: a retrospective cross-sectional real-world study. Diabetologia. 2024 Aug;67(8):1527-1535. doi: 10.1007/s00125-024-06171-y. Epub 2024 May 24. PMID 38787436
- [Derived] De Ridder F, Charleer S, Jacobs S, Bolsens N, Ledeganck KJ, Van Aken S, Vanbesien J, Gies I, Casteels K, Massa G, Lysy PA, Logghe K, Lebrethon MC, Depoorter S, Gillard P, De Block C, den Brinker M. Effect of nationwide reimbursement of real-time continuous glucose monitoring on HbA1c, hypoglycemia and quality of life in a pediatric type 1 diabetes population: The RESCUE-pediatrics study. Front Pediatr. 2022 Oct 6;10:991633. doi: 10.3389/fped.2022.991633. eCollection 2022. PMID 36275049
- [Derived] Charleer S, De Block C, Nobels F, Radermecker RP, Lowyck I, Mullens A, Scarniere D, Spincemaille K, Strivay M, Weber E, Taes Y, Vercammen C, Keymeulen B, Mathieu C, Gillard P; RESCUE Trial Investigators. Sustained Impact of Real-time Continuous Glucose Monitoring in Adults With Type 1 Diabetes on Insulin Pump Therapy: Results After the 24-Month RESCUE Study. Diabetes Care. 2020 Dec;43(12):3016-3023. doi: 10.2337/dc20-1531. Epub 2020 Oct 16. PMID 33067260
- [Derived] Charleer S, Mathieu C, Nobels F, De Block C, Radermecker RP, Hermans MP, Taes Y, Vercammen C, T'Sjoen G, Crenier L, Fieuws S, Keymeulen B, Gillard P; RESCUE Trial Investigators. Effect of Continuous Glucose Monitoring on Glycemic Control, Acute Admissions, and Quality of Life: A Real-World Study. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1224-1232. doi: 10.1210/jc.2017-02498. PMID 29342264